CLINICAL TRIAL: NCT01376622
Title: Changes in Pituitary Iron and Volume With Deferasirox in Transfusional Iron Overload
Brief Title: Changes in Pituitary Iron and Volume With Deferasirox
Status: Completed | Type: Observational
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, John C. Wood, Principal Investigator, Children's Hospital Los Angeles
Other Study IDs: CCI-08-00143
Record Dates: First submitted 2011-06-17; First posted 2011-06-20 (Estimated); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Iron Overload
MeSH Terms: conditions — Iron Overload

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronically Transfusion Patients: Patients with transfusion dependent anemia (excluding sickle cell disease), ages 2-25, on Deferasirox chelation therapy, to be monitored over 2 years.
- Controls: Normal controls, ages 2-25, with no known brain abnormality or endocrine dysfunction.

SUMMARY:
Despite continuing advances in iron chelation therapy, iron toxicity of endocrine glands, particularly the pituitary gland, remains common in patients with transfusion dependent anemias. We would like to establish accurate population norms of pituitary R2 and volume and understand the progression of pituitary iron in transfused patients on Deferasirox.

ELIGIBILITY:
Inclusion Criteria:

* Currently on chronic transfusion therapy.
* Duration of chronic transfusion >1 year.
* Age 2 to 25 years
* On deferasirox monotherapy for the duration of the study.
* Informed consent from legal guardian and/or patient.
* On deferasirox for a minimum of 3 months at start of study.

Exclusion Criteria:

* Sickle cell disease or sickle-beta zero genotype.
* Combination of deferasirox and another iron chelator.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Transfusion Dependent Anemia
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2008-11; Primary Completion 2011-07-01 (Actual); Study Completion 2011-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C Wood, MD, PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Result] Wood JC, Noetzl L, Hyderi A, Joukar M, Coates T, Mittelman S. Predicting pituitary iron and endocrine dysfunction. Ann N Y Acad Sci. 2010 Aug;1202:123-8. doi: 10.1111/j.1749-6632.2010.05545.x. PMID 20712782